CLINICAL TRIAL: NCT06299150
Title: Clinical Evaluation of Three Different Techniques Restoring Ellis Class II Traumatized Central Incisors In Children: Randomized Clinical Trial
Brief Title: Clinical Evaluation of Three Different Techniques Restoring Ellis Class II Traumatized Central Incisors In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Salmoon, Principal Investigator, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1
Record Dates: First submitted 2024-02-23; First posted 2024-03-07 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Composites Resins
MeSH Terms: interventions — IPS e.max CAD LT

STUDY DESIGN:
Intervention Model Description: The study is a randomized clinical trial (RCT) where 2 arm parallel groups with a 1:1 allocation ratio were compared. The child participants and the legal guardian of each participating child and the statistician were blinded.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct resin composite mini-veneer (Active Comparator): Composites resins have become the first choice for direct anterior and posterior restorations. The great popularity is related to their esthetic appearance and reduced need of sound tissue removal as compared with former treatments. Several studies have demonstrated that composite restorations may last long in clinical service. Composite restorations have demonstrated a good clinical performance with annual failure rates varying from 1% to 3% in posterior teeth and 1% to 5% in anterior teeth.
  Interventions: Other: IPS e.max CAD
- IPS e.max CAD (Experimental): "IPS e max" likely refers to a type of dental material or technology. IPS e.max is a popular brand of lithium disilicate glass-ceramic used in dentistry for the fabrication of dental restorations such as crowns, veneers, inlays, onlays, and bridges.
  IPS e.max restorations are known for their excellent esthetics, strength, and durability. They are designed to closely mimic the natural appearance of teeth while providing reliable performance and longevity. Dentists often choose IPS e.max restorations for their patients due to their versatility and ability to meet both esthetic and functional requirements.
  Interventions: Other: IPS e.max CAD

INTERVENTIONS:
Other: IPS e.max CAD — CAD CAM Restoration

SUMMARY:
Dental trauma (DT) of the incisors and their supporting tissues, one of the most challenging dental emergencies, requires immediate assessment and management due to psychological and physical reasons. This is especially important for young permanent teeth to minimize undesired complications. The treatment of dental trauma is sometimes neglected, although it might lead to pain, difficulty in articulation and mastication, and considerable negative effects on a patient's self-esteem. However, the aesthetics of the anterior teeth are very important aspects of human appearance and can be affected by many factors, including the presence of fillings, tooth color, position, alignment, shape, and number.

Rasmussen ST et al. discovered in 1981 that most children suffer from tooth trauma. According to their research, 25% of all schoolchildren and 33% of adults have undergone trauma, with the majority of cases occurring before the age of 19.

As the maxillary incisors are the most commonly injured teeth due to their exposed position, a functional, aesthetic, and time-efficient restoration is frequently demanded. According to the current International Association of Dental Traumatology guidelines, crown fractures confined to enamel and dentine may be treated either with a direct composite restoration or with an adhesive reattachment of the fractured fragment. As long as the fragment is intact, reattachment is often preferred in dental practice. This technique facilitates the restoration of the tooth with its original anatomy, color, and function in a minimum amount of time. Unfortunately, clinical studies regarding the survival of reattached fragments are scarce, and results from laboratory investigations cannot be transferred to clinical settings without limitations. Furthermore, longevity data of direct composite restorations in fractured anterior teeth are restricted to a few clinical studies.

In addition to the aforementioned restorative alternatives, the use of small partial glassy restorations-partial laminate veneers (PLVs), sectional veneers, or ceramic fragments has become increasingly popular over the last few years. PLVs are thin pieces of glass matrix ceramic fragments without a defined shape that are used to restore small defects in the anterior teeth. As tooth preparation is not required for this type of restoration, and minimal to no prep is accepted, the maximum amount of enamel surface structure is conserved. Thus, retention relies completely on adhesion, which is primarily achieved by bonding to the conditioned glassy surface. Despite their growing popularity, available data in the literature on PLVs are limited to a few in vitro studies and case reports, without any clinical information available at present.

Patients in all groups will receive a minimally invasive restoration with high esthetic advantages and long-term success of their fractured incisors (either conventional composite restoration, fragment reattachment, or partial laminate veneers) that require minimal to no preparation and do not require local anesthesia.

DETAILED DESCRIPTION:
Aim of the study:

This randomized clinical trial study will assess the survival and success rates of three different types of conservative restorations restored the Ellis Class II traumatized central incisors by clinical evaluation of the patients.

Research question:

Are the direct resin composite mini-veneer, reattachment of broken segments and IPS e.max CAD clinically successful techniques in restoring Ellis Class II traumatized central incisors in children?

PICOS:

P: Patients above 8 years old with traumatized upper incisor I (1): Partial laminate veneers (PLV) I (2): Fragment reattachment C: Conventional composite restoration O: Clinical Success S: In-Vivo Study

II. Methods

Study Design:

Study Type: Interventional (Clinical Trial) Estimated Enrolment: 40 participants Allocation: Randomized Intervention Model: Parallel Assignment Primary Purpose: Treatment Official Title: Clinical Evaluation of Three Different Techniques restoring

Ellis Class II traumatized central incisors in children:

Randomized Clinical Trial Estimated Study Start Date: December 2023 Estimated Primary Completion Date: January 2024

Trial design:

The study is a randomized clinical trial (RCT) where 2 arm parallel groups with a 1:1 allocation ratio were compared. The child participants and the legal guardian of each participating child and the statistician were blinded.

Outcome Measures:

1. Primary outcome: Clinical success/ survival [Time Frame: 12 months].

   * Clinical success will evaluate using (a modified version of the United States Public Health Service (USPHS) criteria). [Appendix A]
   * Each parameter will assess using visual and tactile observations (probe and mirror).
   * At the checkup visits (3, 6, 9, 12 months), will take standardized photographs and the restorations will clinically evaluate by an independent and calibrated clinician.
   * The need for replacement and partial fractures (chippings) will define as failures
2. Secondary outcomes: [Time Frame: 12 months].

   * Marginal adaptation: using Trios 3 scanner via scan compare (microns)
   * Colour change: using Trios 3 scanner via scan compare (yes or no binary)
   * Patient centred outcomes to the restoration: Patient's satisfaction questioner. (33) [Appendix B] Eligibility Criteria

Ages Eligible for Study: 8 - 18 Years Sexes Eligible for Study: All Accepts Healthy Volunteers: Yes

Criteria

Inclusion Criteria:

1. 8-18 years old
2. Ellis Class II traumatized central incisors
3. Controlled dental disease - no active caries or periodontal diseases
4. Patients will be available to be clinically reviewed up to 1 year

Exclusion Criteria:

1. All Ellis Classification traumatized central incisors except Ellis Class II
2. Patients with uncontrolled active tooth decay or periodontal disease (i.e. 4+ mm probing depth and bleeding on probing).
3. Poor oral hygiene and motivation.
4. Patients with parafunctional habits (e.g., bruxism, biting on hard objects).
5. Patients with debilitating illnesses or complicating medical conditions

Explanation for choice of comparators:

Composites resins have become the first choice for direct anterior and posterior restorations. The great popularity is related to their esthetic appearance and reduced need of sound tissue removal as compared with former treatments. Several studies have demonstrated that composite restorations may last long in clinical service. Composite restorations have demonstrated a good clinical performance with annual failure rates varying from 1% to 3% in posterior teeth and 1% to 5% in anterior teeth. (34)

Thus, direct resin composites offer several advantages to both patients and clinicians, including a reduction in treatment costs and clinical working times (i.e., fewer clinical appointments), as well as reversibility and reparability of the treatment. For these reasons, most clinicians consider resin composites as the material of choice when maximum preservation of the tooth structure is required. (24,35)

Sample size (Power analysis):

Sample size calculated depending on a previous study (Oosterhaven et al., 2023) as reference. (24) According to this study, the probability of color match (clinical success) in group 1 is 0.98. If the estimated probability of group 2 is 0.6, we will need to study 17 cases in each group with probability (power) 0.8. The Type I error probability. Total sample size increased to 20 subjects per group to compensate for a 15 % drop out during follow up. Sample size calculation was achieved using chi-squared test to evaluate that was performed by using P.S. Power3.1.6, software Version 3.1.2 (Vanderbilt University, Nashville, Tennessee, USA.

Statistical Methods

Statistical analysis:

Data were collected, tabulated, and statistically analyzed using Microsoft Excel ® 2016, Statistical Package for Social Science (SPSS)® Ver. 24. And Minitab ® statistical software Ver. 16.

Handling of numerical / quantitative variables:

Numerical data will be explored for normality by checking the data distribution using Kolmogorov- Smirnov and Shapiro-Wilk tests. Data will be presented as mean & standard deviation. If data will be normally distributed comparison between 2 different groups will be performed by using independent t-test, comparison between 2 related groups will be performed by using Paired t-test, while comparison between more than 2 groups will be performed by using One Way ANOVA test followed by Tukey's Post Hoc test for multiple comparisons. If data will be non-parametric data comparison between 2 different groups will be performed by using Mann-Whitney test, comparison between 2 related groups will be performed by using Wilcoxon Signed Rank test, while comparison between more than 2 groups will be performed by using Kruskal-Walli's test.

Handling of categorial / qualitative variables:

Data will be presented as frequency and percentages. All comparisons will be performed by using Chi square test.

Recruitment:

The study will be conducted at the pediatric dentistry department of MSA University pediatric outpatients. All subjects will be monitored and reviewed every 3 months for 12 months.

Post-trial care

* Oral hygiene instructions and serving brush and toothpaste
* Dietary recommendations

ELIGIBILITY:
Inclusion Criteria:

1. 8-18 years old
2. Ellis Class II traumatized central incisors
3. Controlled dental disease - no active caries or periodontal diseases
4. Patients will be available to be clinically reviewed up to 1 year

Exclusion Criteria:

1. All Ellis Classification traumatized central incisors except Ellis Class II
2. Patients with uncontrolled active tooth decay or periodontal disease (i.e. 4+ mm probing depth and bleeding on probing).
3. Poor oral hygiene and motivation.
4. Patients with parafunctional habits (e.g., bruxism, biting on hard objects).
5. Patients with debilitating illnesses or complicating medical conditions

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical success/ survival | 12 months
  * Clinical success will evaluate using (a modified version of the United States Public Health Service (USPHS) criteria). [Appendix A]
  * Each parameter will assess using visual and tactile observations (probe and mirror).
  * At the checkup visits (3, 6, 9, 12 months), will take standardized photographs and the restorations will clinically evaluate by an independent and calibrated clinician.
  * The need for replacement and partial fractures (chippings) will define as failures

CONTACTS AND LOCATIONS:
Locations (1):
- MSA University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No